CLINICAL TRIAL: NCT04990362
Title: Effects of Pomegranate Seed Oil and Mediterranean Diet at Motor Skills and Cognitive Abilities in Mild Cognitive Impairment.
Brief Title: Effects of Pomegranate Seed Oil and Mediterranean Diet on MCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Greek Alzheimer's Association and Related Disorders (Other)
Responsible Party: Principal Investigator, Magda Tsolaki, Professor of Neurology, Medical School, Aristotle University of Thessaloniki Affiliation: Aristotle University of Thessaloniki, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 69/5-6-2021
Record Dates: First submitted 2021-07-26; First posted 2021-08-04 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Cognition; Mental Health; APOE; ε3/ε3; ε3/ε2; ε3/ε4; ε2/ε4; ε4/ε4; Pomegranate oil
MeSH Terms: conditions — Cognitive Dysfunction; Psychological Well-Being | interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MD + Seed oil (Experimental): Pomegranate oil + Mediterranean Diet 30 patients Mediterranean dietary protocol Dietary Supplement: Pomegranate oil in a glass bottle of 30ml Dietary Supplement: Mediterranean dietary protocol
  Intervention:
  Mediterranean diet, Pomegranate oil
  Interventions: Dietary Supplement: Pomegranate oil, Mediterranean Diet
- MD (Active Comparator): Mediterranean Diet 30 patients Mediterranean dietary protocol Dietary Supplement: Mediterranean dietary protocol Intervention: Mediterranean diet
  Interventions: Dietary Supplement: Mediterranean Diet

INTERVENTIONS:
Dietary Supplement: Pomegranate oil, Mediterranean Diet — Dietary Supplement: Pomegranate oil in a glass bottle of 0.15ml per day +Mediterranean dietary protocol Dietary Supplement: Mediterranean dietary protocol
  Arms: MD + Seed oil
Dietary Supplement: Mediterranean Diet — Dietary Supplement: Mediterranean dietary protocol
  Arms: MD

SUMMARY:
A double-blind clinical trial of pomegranate oil and Mediterranean diet that will be carried out on 60 patients with Mild Cognitive Impairment (MCI) and APOE ε3 and ε4 allele.

The aim of the research is to examine if the Mediterranean diet with pomegranate oil and without it can bring positive changes in patients with MCI in terms of motor and cognitive skills.

DETAILED DESCRIPTION:
OBJECTIVES OF THE TRIAL

The objectives of this study are:

To investigate the efficacy of Mediterranean diet and Pomegranate oil as a disease course modifying treatment for MCI.

STUDY DESIGN This is a Greek, controlled double-blind trial of two compared groups, one with Mediterranean diet and one with Mediterranean diet and pomegranate oil. Qualifying patients will be assigned to receive 0.15 mL of pomegranate oil every day with Mediterranean diet at one group and at the other group will not. A Mediterranean dietary protocol will be given on a daily basis for 12 months at both groups.

Duration The total study duration will be 12 months. The recruitment will be about 6 months and the statistics and the preparation of the paper other 6 months.

Number of Subjects:

Sixty (60) subjects total will be enrolled.; Thirty (30) in the A group (Pomegranate oil + Mediterranean Diet); Thirty (30) in the B Group (Mediterranean Diet).

Patient identification:

Initials (First initial of first name and First initial of surname), date of birth and Patient Identification Number from database empedocles.

Eligibility Screening Form (ESF) : Checklist of inclusion and exclusion criteria Eligibility Statement: for patients found to be ineligible, the reason for ineligibility must be stated and Written informed consent will be obtained from the subjects which are eligible. The informed consent form must be co-signed by the physician. The nature of the study and the potential risks associated with the trial will be explained to all subjects- candidates and their responsible informants.

Signature and date: the ESF may be completed by a research assistant but it is required that the principal investigator/study clinician sign and date the ESF to verify eligibility of the patient for inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Mild Cognitive Impairment
* Carry APOE ε3 or ε4 genes

Exclusion Criteria:

* Diagnosis of Dementia
* Patients who receive medication for memory or depression
* Patients who do not carry APOE ε3 or ε4 genes

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination (MMSE | baseline,12 months
  Score scale:0-30,cut off:24
FUCAS | baseline,12 months
  Measurements to Assess Daily Functionality Changes in Functional cognitive assessment scale (FUCAS) score Score scale:42-126,cut off:42
Letter & Category Fluency Test | baseline,12 months
  Measurement to Assess Verbal Fluency and Learning Changes in the Letter & Category Fluency Test
CDR | baseline,12 months
  Measurements to Assess General Cognitive Function Changes in Global Clinical Dementia Rating (CDR)
MoCA | baseline,12 months
  Measurements to Assess General Cognitive Function Changes in Montreal Cognitive Assessment (MoCA)
CANTAB | baseline,12 months
  Measurements to Assess General Cognitive Function Changes in Cambridge Neuropsychological Test Automated Battery (CANTAB)
Clock Drawing test | baseline,12 months
  Measurements to Assess General Cognitive Function Changes in the Clock Drawing test
Logical Memory test | baseline,12 months
  Measurements to Assess General Cognitive Function Changes in the Logical Memory test
Digit Span Forward & Backward test | baseline,12 months
  Measurements to Assess General Cognitive Function Changes in the Digit Span Forward & Backward test
WAIS-R Digit Symbol | baseline,12 months
  Measurements to Assess General Cognitive Function Changes in the WAIS-R Digit Symbol Substitution Test
TMT part A and B | baseline,12 months
  Measurements to Assess General Cognitive Function Changes in the Trail Making Test
ADASCog | baseline,12 months
  Measurements to Assess Daily Functionality Changes in Alzheimer's Disease Assessment Scale-Cognitive (ADASCog)
Functional Rating Scale for Dementia | baseline,12 months
  Measurements to Assess Daily Functionality Changes in Functional Rating Scale for Dementia (FRSSD)
Auditory Verbal Learning Test | baseline,12 months
  Measurement to Assess Verbal Fluency and Learning Changes in the Auditory Verbal Learning Test
Boston Naming Test | baseline,12 months
  Measurement to Assess Verbal Fluency and Learning Changes in the Boston Naming Test
Fullerton Functional Test | baseline,12 months
  Measurement to Assess Physical Abilities

CONTACTS AND LOCATIONS:
Overall Officials: Magda Tsolaki, MD PhD Prof., Study Chair — Greek Alzheimer's Association and Related Disorders; Thanos Chatzikostopoulos, MSc, Principal Investigator — Greek Alzheimer's Association and Related Disorders
Locations (1):
- Alzheimer Hellas, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No
Participants' personal data will not be shared with other researchers